CLINICAL TRIAL: NCT04039295
Title: Estimation of Injection Volume for Caudal Epidural Block Using Dynamic Ultrasound Imaging in Young Pediatric Patients: an Observational Study
Brief Title: Estimation of Injection Volume for Caudal Epidural Block Using Dynamic US Imaging in Children
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Hajung Kim, Clinical instructor, Asan Medical Center
Other Study IDs: 2019-0750
Record Dates: First submitted 2019-07-24; First posted 2019-07-31 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Caudal Epidural Block

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: ultrasound guided caudal epidural block — dynamic ultrasound imaging of the spread of local anesthetics

SUMMARY:
Caudal epidural block is the most commonly used technique for analgesia in pediatric patients. Although there are clinically used doses of local anesthetics for caudal epidural block, we do not know exactly how much levels are blocked in young children. Thus, we aimed to identify the spreading of injection of local anesthetics for caudal epidural block using ultrasound imaging in young children.

ELIGIBILITY:
Inclusion Criteria:

* age: 6-24months
* ASA 1-3
* body weight: 5-20kg

Exclusion Criteria:

* patients who refuse to participate
* local site infection, pilonidal cyst, spina bifida
* spinal/meningeal abnormality
* patients who discharge after surgery without admission
* patients who is judged ineligible for other reasons by the authors

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Among the patients who are scheduled to undergo elective polydactyly / syndactyly / polysyndactyly correction surgery in Asan Medical Center, the patients who meet the inclusion criteria are included.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-14 (Actual)

PRIMARY OUTCOMES:
Required volume of local anesthetics | 1 day
  Required volume of local anesthetics to reach each level

CONTACTS AND LOCATIONS:
Overall Officials: Hyungtae Kim, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim HJ, Kim H, Lee S, Koh WU, Park SS, Ro Y. Reconsidering injection volume for caudal epidural block in young pediatric patients: a dynamic flow tracking experimental study. Reg Anesth Pain Med. 2024 May 7;49(5):355-360. doi: 10.1136/rapm-2023-104409. PMID 37429622